CLINICAL TRIAL: NCT00298831
Title: A Multicenter, Open Label, Phase IIIa Trial to Evaluate the Efficacy and Safety of Org 25969 When Used at the End of a Surgical Procedure to Reverse the Neuromuscular Block Induced by Rocuronium Following Routine Anesthesia
Brief Title: Use of Sugammadex at the End of Case in Routine Anesthesia (MK-8616-023)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05943; 19.4.311 (Other: Organon Protocol Number); P05943 (Other: Schering-Plough Protocol Number); MK-8616-023 (Other: Merck Protocol Number)
Record Dates: First submitted 2006-03-01; First posted 2006-03-03 (Estimated); Results first posted 2019-03-15 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Anesthesia, General
MeSH Terms: interventions — Sugammadex; Rocuronium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sugammadex (Experimental): Each participant received an intravenous single bolus dose of 0.6 mg/kg rocuronium. If further neuromuscular block was required after endotracheal intubation, maintenance dose(s) of 0.15 mg/kg rocuronium was administered. At least 15 minutes after the intubation dose or the last maintenance dose of rocuronium, an intravenous single bolus dose of 4.0 mg/kg MK-8616 was administered.
  Interventions: Drug: Sugammadex; Drug: Rocuronium

INTERVENTIONS:
Drug: Sugammadex — At least 15 minutes after the intubation dose or the last maintenance dose of rocuronium, an intravenous single bolus dose of 4.0 mg/kg Org 25969 was administered.
  Other Names: Org 25969; MK-8616
Drug: Rocuronium — Each participant received an intravenous single bolus dose of 0.6 mg/kg rocuronium. If further neuromuscular block was required after endotracheal intubation, maintenance dose(s) of 0.15 mg/kg rocuronium was/were administered.

SUMMARY:
The primary purpose of the study is to determine the time-course of recovery to a T4/T1 ratio of 0.9 within 4 minutes after 4.0 mg.kg^-1 Sugammadex is administered at least 15 minutes after the last administration of rocuronium in a wide range of surgical procedures and anesthetic regimens (routine use). Safety evaluation is part of the study.

ELIGIBILITY:
Inclusion criteria:

* American Society of Anesthesiologists (ASA) Class 1-3 participants who are scheduled to undergo an elective surgical procedure under general anesthesia requiring neuromuscular relaxation with the use of rocuronium.

Exclusion criteria:

* Participants with neuromuscular disorders, significant renal dysfunction, malignant hyperthermia, allergy to medications used in general anesthesia and in whom difficult intubation is expected.
* Participants taking medications known to interfere with neuromuscular blocking agents.
* Participants who are of child-bearing potential, pregnant, and breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2005-10-27 (Actual); Primary Completion 2006-05-22 (Actual); Study Completion 2006-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Hudson ME, Rietbergen H, Chelly JE. Sugammadex is effective in reversing rocuronium in the presence of antibiotics. BMC Anesthesiol. 2014 Aug 15;14:69. doi: 10.1186/1471-2253-14-69. eCollection 2014. PMID 25157214
- See also: Click here to access a synopsis of the study results. — http://www.merck.com/clinical-trials/policies-perspectives.html
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in 19 trial sites in the United States.
Period: Overall Study
Arm/Group | Sugammadex
Started | 224
Treated | 197
Completed | 192
Not Completed | 32
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 1
Not completed — Participants did not receive treatment | 27

BASELINE CHARACTERISTICS:
Population: The analysis population was all randomized and treated participants.
Arm/Group | Sugammadex
Number analyzed (Participants) | 197
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The analysis population was all randomized and treated participants.
  Years | 53 (15)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The analysis population was all randomized and treated participants.
  Participants
    Female | 103
    Male | 94
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The analysis population was all randomized and treated participants.
  Participants
    American Indian or Alaska Native | 0
    Asian | 5
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 18
    White | 172
    More than one race | 0
    Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Time From Start of MK-8616 Administration to Recovery of the T4/T1 Ratio to 0.9
Description: Mean time from start of MK-8616 administration to recovery of participant T4/T1 ratio to 0.9 was assessed through the repeated application (every 15 seconds) of an electrical stimulation protocol. Specifically, 4 electrical stimulations were applied to the ulnar nerve and the magnitude of the twitch response of the adductor pollicis muscle (i.e. thumb twitch response) was assessed. With T4 and T1 referring to the respective magnitude of the fourth and first thumb twitch during nerve stimulation, the T4/T1 ratio indicates the current degree of neuromuscular blockade (NMB) present in the participant as a decimal from 0 (loss of T4 twitch) to 1 (no NMB). Further, reduced recovery time of the T4/T1 ratio to 0.9 indicates faster recovery from NMB. Summary data, originally presented in the format of units "minutes:seconds" (mm:ss), was reformatted to be presented in the single unit of "minutes" (min).
Time Frame: Up to approximately 30 minutes following administration of study treatment
Population: The analysis population consisted of all treated participants had at least one post baseline T4/T1 ratio to 0.9 efficacy measurement.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Sugammadex
Number analyzed (Participants) | 177
Minutes | 2.32 (2.15)

2. Secondary Outcome: Time From Start of MK-8616 Administration to Recovery of the T4/T1 Ratio to 0.7
Description: Mean time from start of MK-8616 administration to recovery of participant T4/T1 ratio to 0.7 was assessed through the repeated application (every 15 seconds) of an electrical stimulation protocol. Specifically, 4 electrical stimulations were applied to the ulnar nerve and the magnitude of the twitch response of the adductor pollicis muscle (i.e. thumb twitch response) was assessed. With T4 and T1 referring to the respective magnitude of the fourth and first thumb twitch during nerve stimulation, the T4/T1 ratio indicates the current degree of neuromuscular blockade (NMB) present in the participant as a decimal from 0 (loss of T4 twitch) to 1 (no NMB). Further, reduced recovery time of the T4/T1 ratio to 0.7 indicates faster recovery from NMB. Summary data, originally presented in the format of units "minutes:seconds" (mm:ss), was reformatted to be presented in the single unit of "minutes" (min).
Time Frame: Up to approximately 10 minutes following administration of study treatment
Population: The analysis population consisted of all treated participants had at least one post baseline T4/T1 ratio to 0.7 efficacy measurement.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Sugammadex
Number analyzed (Participants) | 188
Minutes | 1.50 (1.07)

3. Secondary Outcome: Time From Start of MK-8616 Administration to Recovery of the T4/T1 Ratio to 0.8
Description: Mean time from start of MK-8616 administration to recovery of participant T4/T1 ratio to 0.8 was assessed through the repeated application (every 15 seconds) of an electrical stimulation protocol. Specifically, 4 electrical stimulations were applied to the ulnar nerve and the magnitude of the twitch response of the adductor pollicis muscle (i.e. thumb twitch response) was assessed. With T4 and T1 referring to the respective magnitude of the fourth and first thumb twitch during nerve stimulation, the T4/T1 ratio indicates the current degree of neuromuscular blockade (NMB) present in the participant as a decimal from 0 (loss of T4 twitch) to 1 (no NMB). Further, reduced recovery time of the T4/T1 ratio to 0.8 indicates faster recovery from NMB. Summary data, originally presented in the format of units "minutes:seconds" (mm:ss), was reformatted to be presented in the single unit of "minutes" (min).
Time Frame: Up to approximately 15 minutes following administration of study treatment
Population: The analysis population consisted of all treated participants had at least one post baseline T4/T1 ratio to 0.8 efficacy measurement.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Sugammadex
Number analyzed (Participants) | 188
Minutes | 1.80 (1.37)

4. Secondary Outcome: Clinical Assessment of Recovery - Participant's Level of Consciousness
Description: The quality of recovery was assessed by asking the participant 40 questions from a validated Quality of Recovery Questionnaire (QoR-40). Participants were assessed for level of consciousness (i.e., awake and oriented, arousable with minimal stimulation, responsive only to tactile stimulation), if applicable, by asking their name, if they are aware of where they are, and what day it is. Assessment 1 occurred prior to transfer to the recovery room after extubation and Assessment 2 occurred prior to discharge from the recovery room.
Time Frame: Up to 24 hours
Population: The analysis population consisted of all participants who received investigational product and had at least one post baseline efficacy measurement for the analysis endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Sugammadex
Number analyzed (Participants) | 197
Participants
  Awake and oriented - Assessment 1 | 138
  Awake and oriented - Assessment 2 | 184
  Arousable with minimal stimulation - Assessment 1 | 51
  Arousable with minimal stimulation - Assessment 2 | 12
  Responsive only to tactile stimulation - Assess. 1 | 8
  Responsive only to tactile stimulation - Assess. 2 | 0

5. Secondary Outcome: Clinical Assessments of Recovery - Participant Able to Perform 5-second Head Lift (5SHL)
Description: 5-second head lift test was assessment of the ability of the participant to lift the head for 5 seconds and was performed by a blinded safety assessor. Tests were repeated every 15 minutes until the participant could successfully perform the 5-second head-lift. Assessment 1 occurred prior to transfer to the recovery room after extubation and Assessment 2 occurred prior to discharge from the recovery room.
Time Frame: Up to 24 hours
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Sugammadex
Number analyzed (Participants) | 197
Participants
  Able to perform 5SHL during Assessment 1 | 173
  Able to perform 5SHL during Assessment 2 | 196

6. Secondary Outcome: Clinical Assessments of Recovery - Check for General Muscle Weakness (GMW)
Description: General muscle weakness check was assessed by the investigator. The assessment of general muscle weakness was based on a scale from 0-10, with 0 representing total paralysis, 1 signifying extreme impairment, 9 for close to no impairment, and 10 for normal muscle strength. Scores of 3, 4, 5, etc. denoted increasing muscle strength in approximately 10% increments. Scores of 9 and lower were denoted as GMW. Assessment 1 occurred prior to transfer to the recovery room after extubation and assessment 2 occurred prior to discharge from the recovery room.
Time Frame: Up to 24 hours
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Sugammadex
Number analyzed (Participants) | 197
Participants
  GMW present during Assessment 1 | 4
  GMW present during Assessment 2 | 9

ADVERSE EVENTS:
Time Frame: Up to 7 days after study drug administration
Description: An adverse event is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study. The population analyzed consisted of all participants who received a dose of the investigational product.
Arm/Group | Sugammadex
All-Cause Mortality (participants affected / at risk) | 0/197
Serious Adverse Events (participants affected / at risk) | 8/197
Other Adverse Events (participants affected / at risk) | 187/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex (N=197)
Electromechanical dissociation (Cardiac disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Peroneal nerve injury (Injury, poisoning and procedural complications) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Radiculitis brachial (Nervous system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Psychiatric symptom (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugammadex (N=197)
Anaemia (Blood and lymphatic system disorders) | 10 (10)
Constipation (Gastrointestinal disorders) | 19 (19)
Nausea (Gastrointestinal disorders) | 77 (80)
Vomiting (Gastrointestinal disorders) | 26 (27)
Chills (General disorders) | 16 (18)
Pyrexia (General disorders) | 25 (25)
Incision site complication (Injury, poisoning and procedural complications) | 23 (24)
Procedural hypertension (Injury, poisoning and procedural complications) | 13 (15)
Procedural hypotension (Injury, poisoning and procedural complications) | 11 (13)
Procedural pain (Injury, poisoning and procedural complications) | 159 (164)
Neutrophil count increased (Investigations) | 10 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (20)
Dizziness (Nervous system disorders) | 27 (29)
Headache (Nervous system disorders) | 25 (27)
Anxiety (Psychiatric disorders) | 10 (10)
Insomnia (Psychiatric disorders) | 20 (20)
Bladder spasm (Renal and urinary disorders) | 12 (12)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 18 (18)
Pruritus (Skin and subcutaneous tissue disorders) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor recognizes the right of the investigator(s) to publish, but all publications must be based on data validated and released by sponsor. Any such scientific paper, presentation, or other communication concerning the clinical trial described in the protocol will first be submitted to sponsor, at least six weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably.